CLINICAL TRIAL: NCT04488588
Title: Survival and 30-days Hospital Outcome in Hospitalized COVID-19 Patients in Upper Egypt: Multi-center Study
Brief Title: Survival and 30-days Hospital Outcome in COVID-19 Patients in Upper Egypt
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU17
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Coronavirus Disease; SARS-CoV-2
Keywords: COVID-19; Survival; 30- Days Hospital outcome; outcome
MeSH Terms: conditions — COVID-19 | interventions — Kaplan-Meier Estimate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kaplan Meier analysis — Kaplan Meier survival analysis was conducted to calculate the cumulative overall survival rates using Log Rank test for comparison between age groups

SUMMARY:
Through history, there have been plenty of pandemics however; the social response to corona virus disease (COVID-19) is unparalleled. It is assessed that almost four billion individuals are living in social segregation during this mother of all pandemics.

Initially described in China in December 2019, severe acute respiratory syndrome caused by corona virus 2 (SARS-CoV-2) has spread all over the world and by 18th July 2020- there was an emergent figure of 13,824,739 confirmed cases and 591.666 losses reported to the WHO. To date, Egypt reported slightly over 82,000 confirmed COVID-19 cases with 3858 deaths. The new pandemic is injuring not only health organizations of several countries but also the financial prudence universal.

Defining the clinical features and associated outcomes of patients diagnosed with coronavirus disease (COVID-19) is fundamental to improving our understanding and adequate management of this illness. Several articles have recently been published, describing the clinical features and outcomes of retrospective individuals with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* This study included 1064 patients consecutively admitted to isolation hospitals in Upper Egypt during the period from 22 March to 23 June 2020

Exclusion Criteria:

* only hospitalized confirmed cases of COVID-19 were included.

Ages: 36 Years to 63 Years | Sex: All
Age Groups: Adult
Study Population: All cases had confirmed COVID-19 infection (based on PCR, chest HRCT, CBC, CRP, Ferritin levels) and received standardized treatment protocols of Ministry of Health and Population based on disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 1064 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
number of co-morbidities in hospitalized patients with COVID-19 | one month
  Determinants of survival in studied covid-19 patients admitted to hospitals
causes of ICU admission | one month
  Determinants of ICU admission in hospitalized patients with COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, MD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - AssiutU, Asyut
  - Aliae Mohamed-Hussein, Asyut

IPD SHARING:
Plan to Share IPD: Undecided